CLINICAL TRIAL: NCT02011945
Title: A Phase 1B Dose Escalation Study to Investigate the Safety, Tolerability and Preliminary Efficacy for the Combination Dasatinib (BMS-354825) Plus Nivolumab (BMS-936558) in Patients Chronic Myeloid Leukemia (CML)
Brief Title: A Phase 1B Study to Investigate the Safety and Preliminary Efficacy for the Combination of Dasatinib Plus Nivolumab in Patients With Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-373; 2013-002156-33 (EudraCT Number)
Record Dates: First submitted 2013-11-21; First posted 2013-12-16 (Estimated); Results first posted 2019-01-17 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-02

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- dasatinib Only (Experimental): dasatinib 100 mg QD(CP) or 140 mg QD (AP)
  Interventions: Drug: Dasatinib
- Dose Level 1 (Experimental): Nivolumab 1 mg/kg q 2 weeks + dasatinib 100 mg QD (CP) or 140 mg QD (AP)
  Interventions: Drug: Dasatinib; Drug: Nivolumab
- Dose Level 2 (Experimental): Nivolumab 3 mg/kg q 2 weeks + dasatinib 100 mg QD (CP) or 140 mg QD (AP)
  Interventions: Drug: Dasatinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Dasatinib
  Other Names: BMS-354825
Drug: Nivolumab
  Other Names: BMS-936558
  Arms: Dose Level 1; Dose Level 2

SUMMARY:
The purpose of this study is to find a dose of Nivolumab that can be safely added to Dasatinib in patients with Chronic Myeloid Leukemia.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Confirmed diagnosis of Chronic Myeloid Leukemia in Chronic Phase or Accelerated Phase :

  * With historically documented Ph+ cells
  * ≥2 prior Tyrosine Kinase Inhibitors (TKI) therapies for CML
  * Currently progressing, resistance to or with a suboptimal response to their most recent therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) Score 0 - 1

Exclusion Criteria:

* Blast phase CML
* Known Abl-kinase mutation resistant to Dasatinib (e.g. T315I or T315A)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-02-07 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- United States (5):
  - Winship Cancer Institute, Atlanta, Georgia
  - Dana Farber Cancer Institute., Boston, Massachusetts
  - Ut Southwestern Medical Center At Dallas, Dallas, Texas
  - The University Of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Local Institution, St Leonards, New South Wales
  - Local Institution, Adelaide, South Australia
  - Local Institution, Parkville, Victoria
- Canada (3):
  - QEII Health Sciences Centre-VG Site, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
- Local Institution, Bordeaux, France
- Germany (4):
  - Campus Virchow Klinikum Der Charite, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinik Frankfurt, Frankfurt am Main
- Italy (3):
  - Local Institution, Napoli
  - Local Institution, Orbassano
  - Local Institution, Roma
- Spain (2):
  - Local Institution, Madrid
  - Local Institution, Valencia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 Participants enrolled; 31 participants randomized. Reasons not randomized: 1 participant withdrew consent, 3 participants no longer met the study criteria.
Period: Overall Study
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Started | 2 | 13 | 16
Completed | 0 | 3 | 6
Not Completed | 2 | 10 | 10
Not completed — Participant requested to Discontinue | 0 | 1 | 1
Not completed — Adverse Event unrelated to Drug | 0 | 2 | 1
Not completed — Study Drug Toxicity | 0 | 0 | 1
Not completed — Treatment Failure | 0 | 7 | 6
Not completed — No Longer Meets Study Criteria | 1 | 0 | 0
Not completed — Proceeded to stem cell transplant | 0 | 0 | 1
Not completed — Sub-Optimal Response to dasatinib | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 2 | 13 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.5 (13.4) | 61.2 (12.4) | 47.1 (13.6) | 53.1 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 5 | 13
  Male | 1 | 6 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 0 | 4 | 8 | 12
  Unknown or Not Reported | 2 | 9 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 4
  White | 2 | 11 | 13 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose Limiting Toxicities (DLT)
Description: DLT will be determined based on the incidence and intensity of drug related adverse events (AEs). The following drug-related AEs (whether related to one or both agents) occurring during the first 6 weeks of combined treatment with both dasatinib plus nivolumab (ie, Weeks 3 to 8, inclusive) would be considered DLTs:
  * Grade 4 hematologic AE lasting > 7 days despite appropriate medical intervention, except as noted below;
  * Grade 3 or Grade 4 nonhematologic AE irrespective of duration;
  * Grade 2 nonhematologic AE lasting > 7 days despite appropriate medical intervention (exception: asymptomatic laboratory values of Grade 2 which do not require medical intervention);
  * Any toxicity managed by discontinuation of nivolumab;
  * Grade ≥ 2 AE not controlled by medical intervention and requiring dasatinib treatment interruption for > 28 consecutive days;
  * Grade ≥ 2 AE not controlled by medical intervention and requiring missing 2 consecutive doses of nivolumab.
Time Frame: Week 3 to week 6
Population: All Treated Participants
Measure: Number; unit: Number of Incidence
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 13 | 16
Number of Incidence | 0 | 0 | 0

2. Primary Outcome: Incidence of Adverse Events (AEs)
Description: Any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational product, whether or not considered related to the investigational product.
Time Frame: Initiation of study drug to discontinuation of nivolumab stop date + 100 days or discontinuation of dasatinib + 30 days
Population: All Treated Participants
Measure: Number; unit: Number of Adverse Events
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 13 | 16
Number of Adverse Events
  CML-CP, No Prior dasatinib treatment: number analyzed (Participants) | 0 | 1 | 2
  CML-CP, No Prior dasatinib treatment |  | 1 | 2
  CML-CP, Prior dasatinib treatment: number analyzed (Participants) | 2 | 8 | 11
  CML-CP, Prior dasatinib treatment | 1 | 8 | 11
  CML-AP participants: number analyzed (Participants) | 0 | 4 | 3
  CML-AP participants |  | 4 | 3

3. Primary Outcome: Incidence of Serious Adverse Events (SAEs)
Description: Any untoward medical occurrence that at any dose: results in death, is life threatening, requires in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is a important medical event.Requires inpatient hospitalization or causes prolongation of existing hospitalization, results.
Time Frame: Initiation of study drug to within 100 days of discontinuation of nivolumab dosing and 30 days of dasatinib dosing
Population: All Treated Participants
Measure: Number; unit: Number of Adverse Events
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 13 | 16
Number of Adverse Events
  CML-CP, No Prior dasatinib treatment: number analyzed (Participants) | 0 | 1 | 2
  CML-CP, No Prior dasatinib treatment |  | 0 | 2
  CML-CP, Prior dasatinib treatment: number analyzed (Participants) | 2 | 8 | 11
  CML-CP, Prior dasatinib treatment | 0 | 3 | 4
  CML-AP participants: number analyzed (Participants) | 0 | 4 | 3
  CML-AP participants |  | 4 | 2

4. Primary Outcome: Incidence of Change From Baseline in Clinical Laboratory Tests: Hematology
Description: The number of participants with a shift in laboratory test results from baseline to Grade 3-4 in hematology
Time Frame: Up to 40 Months
Population: All Treated Participants
Measure: Number; unit: Participants
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 13 | 16
Participants
  Hemoglobin | 0 | 2 | 4
  Platelets | 0 | 5 | 4
  Absolute Neutrophil Count (ANC) | 0 | 5 | 3
  White Blood Cell (WBC) | 0 | 1 | 3

5. Primary Outcome: Incidence of Abnormalities in Clinical Laboratory Tests: Liver Tests
Description: The number of participants with an abnormal Liver function test.
  Aspartate aminotransferase (AST) Alanine aminotransferase (ALT) Upper Limit of Normal (ULN)
Time Frame: Up to 40 Months
Population: All Treated Participants with at least one treatment measure
Measure: Number; unit: Participants
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 13 | 16
Participants
  ALT or AST > 3xULN: number analyzed (Participants) | 1 | 13 | 16
  ALT or AST > 3xULN | 0 | 1 | 1
  ALT or AST > 5xULN: number analyzed (Participants) | 1 | 13 | 16
  ALT or AST > 5xULN | 0 | 0 | 0
  ALT or AST > 10xULN: number analyzed (Participants) | 1 | 13 | 16
  ALT or AST > 10xULN | 0 | 0 | 0
  ALT or AST > 20xULN: number analyzed (Participants) | 1 | 13 | 16
  ALT or AST > 20xULN | 0 | 0 | 0
  Total Bilirubin (Tbili) > 2xULN: number analyzed (Participants) | 1 | 13 | 16
  Total Bilirubin (Tbili) > 2xULN | 0 | 1 | 1
  ALT or AST > 3xULN w/ Tbili > 2xULN within 1 day: number analyzed (Participants) | 1 | 13 | 16
  ALT or AST > 3xULN w/ Tbili > 2xULN within 1 day | 0 | 1 | 0
  ALT or AST > 3xULN w/ Tbili > 2xULN within 30 days: number analyzed (Participants) | 1 | 13 | 16
  ALT or AST > 3xULN w/ Tbili > 2xULN within 30 days | 0 | 1 | 0

6. Primary Outcome: Incidence of Laboratory Abnormalities in Specific Thyroid Tests
Description: Free T3 (FT3) Free T4 (FT4) Lower Limit of Normal (LLN)
Time Frame: Up to 40 Months
Population: All Treated Participants
Measure: Number; unit: Number of Incidences
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 13 | 16
Number of Incidences
  TSH > ULN | 0 | 4 | 4
  TSH > ULN: WITH TSH ≤ ULN AT BASELINE | 0 | 3 | 3
  TSH > ULN: WITH AT LEAST ONE FT3/FT4 TEST < LLN | 0 | 2 | 1
  TSH > ULN: WITH ALL OTHER FT3/FT4 TEST ≥ LLN | 0 | 1 | 1
  TSH > ULN: WITH FT3/FT4 TEST MISSING | 0 | 1 | 2
  TSH > 2*ULN | 0 | 2 | 1
  TSH > 2*ULN: WITH TSH <= ULN AT BASELINE | 0 | 1 | 0
  TSH > 2*ULN: WITH AT LEAST ONE FT3/FT4 TEST < LLN | 0 | 2 | 1
  TSH > 2*ULN: WITH ALL OTHER FT3/FT4 TEST ≥ LLN | 0 | 0 | 0
  TSH > 2*ULN: WITH FT3/FT4 TEST MISSING | 0 | 0 | 0
  TSH < LLN | 0 | 3 | 1
  TSH < LLN: WITH TSH >= LLN AT BASELINE | 0 | 3 | 1
  TSH < LLN: WITH AT LEAST ONE FT3/FT4 TEST > ULN | 0 | 0 | 1
  TSH < LLN: WITH ALL OTHER FT3/FT4 TEST ≤ ULN | 0 | 1 | 0
  TSH < LLN: WITH FT3/FT4 TEST MISSING | 0 | 2 | 0

7. Secondary Outcome: Rate of Major Molecular Response (MMR) : Chronic Myelogenous Leukemia - Chronic Phase (CML-CP), No Prior Dasatinib Participants
Description: Molecular response was assessed using BCR-ABL transcript levels measurement by real-time quantitative polymerase chain reaction (RQ-PCR).
  MMR is defined as ≥ 3-log reduction in BCR-ABL transcripts or a ratio of ≤ 0.1% on the International Scale (IS).
Time Frame: upto 36 Months
Population: All treated Participants, CML-CP no prior Dasatinib participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 1 | 2
Percentage of Participants
  MMR Rate by 6 Months |  | 100 [2.5 to 100] | 0 [0 to 84.2]
  MMR Rate by 12 Months |  | 100 [2.5 to 100] | 0 [0 to 84.2]
  MMR Rate by 24 Months |  | 100 [2.5 to 100] | 0 [0 to 84.2]
  MMR Rate by 36 Months |  | 100 [2.5 to 100] | 0 [0 to 84.2]

8. Secondary Outcome: Rate of Major Molecular Response (MMR) : Chronic Myelogenous Leukemia - Chronic Phase (CML-CP), Prior Dasatinib Participants
Description: as for outcome 7
Time Frame: upto 36 Months
Population: All treated Participants, CML-CP prior Dasatinib participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 8 | 11
Percentage
  MMR Rate by 6 Months | 0 [0 to 84.2] | 25 [3.2 to 65.1] | 18.2 [2.3 to 51.8]
  MMR Rate by 12 Months | 0 [0 to 84.2] | 25 [3.2 to 65.1] | 27.3 [6.0 to 61.0]
  MMR Rate by 24 Months | 0 [0 to 84.2] | 25 [3.2 to 65.1] | 36.4 [10.9 to 69.2]
  MMR Rate by 36 Months | 0 [0 to 84.2] | 25.0 [3.2 to 65.1] | 45.5 [16.7 to 76.6]

9. Secondary Outcome: Rate of Major Molecular Response (MMR) : Chronic Myelogenous Leukemia - Advanced Phase (CML-AP) Participants
Description: as for outcome 7
Time Frame: upto 36 Months
Population: All treated Participants, CML-AP Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 4 | 3
Percentage
  MMR Rate by 6 Months |  | 0 [0.0 to 60.2] | 33.3 [0.8 to 90.6]
  MMR Rate by 12 Months |  | 0 [0.0 to 60.2] | 66.7 [9.4 to 99.2]
  MMR Rate by 24 Months |  | 0 [0.0 to 60.2] | 66.7 [9.4 to 99.2]
  MMR Rate by 36 Months |  | 0 [0.0 to 60.2] | 66.7 [9.4 to 99.2]

10. Secondary Outcome: Rate of Molecular Response 4.5 (MR4.5) : Chronic Myelogenous Leukemia - Chronic Phase (CML-CP), No Prior Dasatinib Participants
Description: Molecular response was assessed using BCR-ABL transcript levels measurement by real-time quantitative polymerase chain reaction (RQ-PCR).
  A molecular response 4.5 (MR4.5) was defined as ≥ 4.5-log reduction in BCR-ABL transcripts or a ratio of ≤ 0.00316% on the International Scale (IS).
Time Frame: upto 36 Months
Population: All treated Participants, CML-CP no prior Dasatinib participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 1 | 2
Percentage
  MR4.5 Rate by 6 Months |  | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 84.2]
  MR4.5 Rate by 12 Months |  | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 84.2]
  MR4.5 Rate by 24 Months |  | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 84.2]
  MR4.5 Rate by 36 Months |  | 100 [2.5 to 100] | 0.0 [0.0 to 84.2]

11. Secondary Outcome: Rate of Molecular Response 4.5 (MR4.5) : Chronic Myelogenous Leukemia - Chronic Phase (CML-CP), Prior Dasatinib Participants
Description: as for outcome 10
Time Frame: upto 36 Months
Population: All treated Participants, CML-CP prior Dasatinib participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 8 | 11
Percentage
  MR4.5 Rate by 6 Months | 0 [0 to 84.2] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5]
  MR4.5 Rate by 12 Months | 0 [0 to 84.2] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5]
  MR4.5 Rate by 24 Months | 0 [0 to 84.2] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5]
  MR4.5 Rate by 36 Months | 0 [0 to 84.2] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5]

12. Secondary Outcome: Rate of Molecular Response 4.5 (MR4.5) : Chronic Myelogenous Leukemia - Advanced Phase (CML-AP) Participants
Description: as for outcome 10
Time Frame: upto 36 Months
Population: All treated Participants, CML-AP Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 4 | 3
Percentage
  MR4.5 Rate by 6 Months |  | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8]
  MR4.5 Rate by 12 Months |  | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8]
  MR4.5 Rate by 24 Months |  | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8]
  MR4.5 Rate by 36 Months |  | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8]

13. Secondary Outcome: Time to Major Molecular Response (MMR) - CML-CP No Prior Dasatinib Participants
Description: measured from the date of first dosing until measurement criteria are first met for MMR. The participants who do not respond will be censored on the date of their last molecular assessment. It is defined for all treated participants.
Time Frame: Up to 36 Months
Population: CML-CP No Prior Dasatinib Subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 1 | 2
Months |  | 0.53 [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

14. Secondary Outcome: Time to Major Molecular Response (MMR) - CML-CP Prior Dasatinib Participants
Description: as for outcome 13
Time Frame: Up to 36 Months
Population: CML-CP Prior Dasatinib participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 8 | 11
Months | NA [NA to NA] — Insufficient number of participants with events | NA [0.56 to NA] — Insufficient number of participants with events | 35.45 [0.95 to NA] — Insufficient number of participants with events

15. Secondary Outcome: Time to Major Molecular Response (MMR) - CML-AP Participants
Description: as for outcome 13
Time Frame: Up to 36 Months
Population: CML-AP Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 4 | 3
Months |  | NA [NA to NA] — Median and Confidence limits not estimable | 5.54 [1.84 to 9.23]

16. Secondary Outcome: Duration of Major Molecular Response (MMR) - CML-CP No Prior Dasatinib Participants
Description: will be computed for participants who have achieved MMR. It will be defined as the time from the first assessment in which MMR, is documented until the first assessment at which disease progression (or confirmed loss of MMR) is documented. Participants who neither progress nor die will be censored on the date of their last molecular assessment
Time Frame: Up to 36 Months
Population: CML-CP No Prior Dasatinib participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 1 | 0
Months |  | NA — Insufficient number of participants with events |

17. Secondary Outcome: Duration of Major Molecular Response (MMR) - CML-CP Prior Dasatinib Participants
Description: as for outcome 16
Time Frame: Up to 36 Months
Population: CML-CP Prior Dasatinib Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 2 | 5
Months |  | NA [23.49 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

18. Secondary Outcome: Duration of Major Molecular Response (MMR) - CML-AP Participants
Description: as for outcome 16
Time Frame: Up to 36 Months
Population: CML-AP Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 0 | 2
Months |  |  | NA [NA to NA] — Insufficient number of participants with events

19. Secondary Outcome: Time to Molecular Response 4.5(MR4.5) - CML-CP No Prior Dasatinib Participants
Description: measured from the date of first dosing until measurement criteria are first met for MR4.5. The participants who do not respond will be censored on the date of their last molecular assessment. It is defined for all treated participants.
Time Frame: Up to 36 Months
Population: CML-CP No Prior Dasatinib Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 1 | 2
Months |  | 35.25 [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

20. Secondary Outcome: Time to Molecular Response 4.5(MR4.5) - CML-CP Prior Dasatinib Participants
Description: as for outcome 19
Time Frame: Up to 36 Months
Population: CML-CP Prior Dasatinib Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 8 | 11
Months | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

21. Secondary Outcome: Time to Molecular Response 4.5(MR4.5) - CML-AP Participants
Description: as for outcome 19
Time Frame: Up to 36 Months
Population: CML-AP Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 4 | 3
Months |  | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

22. Secondary Outcome: Duration of Molecular Response 4.5 (MR4.5) - CML-CP No Prior Dasatinib Participants
Description: will be computed for participants who have achieved MR4.5. It will be defined as the time from the first assessment in which MR4.5, is documented until the first assessment at which disease progression (or confirmed loss of MR4.5 documented. Participants who neither progress nor die will be censored on the date of their last molecular assessment
Time Frame: Up to 36 Months
Population: CML-CP No Prior Dasatinib Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 1 | 0
Months |  | NA — Insufficient number of participants with events |

23. Secondary Outcome: Duration of Molecular Response 4.5 (MR4.5) - CML-CP Prior Dasatinib Participants
Description: as for outcome 22
Time Frame: Up to 36 Months
Population: CML-CP Prior Dasatinib Participants
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Duration of Molecular Response 4.5 (MR4.5) - CML-AP Participants
Description: as for outcome 22
Time Frame: Up to 36 Months
Population: CML-AP Participants
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Initiation of study drug to within 100 days of discontinuation of nivolumab dosing and 30 days of dasatinib dosing
Arm/Group | Dasatinib Only | Dose Level 1 | Dose Level 2
All-Cause Mortality (participants affected / at risk) | 0/2 | 2/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/2 | 7/13 | 8/16
Other Adverse Events (participants affected / at risk) | 1/2 | 13/13 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib Only (N=2) | Dose Level 1 (N=13) | Dose Level 2 (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Device related thrombosis (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib Only (N=2) | Dose Level 1 (N=13) | Dose Level 2 (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 6 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 3
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 6
Vomiting (Gastrointestinal disorders) | 0 | 4 | 6
Asthenia (General disorders) | 0 | 5 | 1
Chest pain (General disorders) | 0 | 2 | 1
Chills (General disorders) | 0 | 1 | 1
Discomfort (General disorders) | 0 | 2 | 0
Face oedema (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 0 | 1 | 3
Mucosal inflammation (General disorders) | 0 | 1 | 1
Oedema (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 2 | 2
Pyrexia (General disorders) | 0 | 5 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 4
Oral herpes (Infections and infestations) | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 2 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Dizziness (Nervous system disorders) | 0 | 3 | 3
Headache (Nervous system disorders) | 0 | 4 | 5
Paraesthesia (Nervous system disorders) | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 1
Dysuria (Renal and urinary disorders) | 0 | 3 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Hot flush (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 1 | 2
Hypotension (Vascular disorders) | 0 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 1
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Implant site pain (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1
Necrosis (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Temperature regulation disorder (General disorders) | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Wound infection bacterial (Infections and infestations) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1
Serum ferritin decreased (Investigations) | 0 | 1 | 0
Spleen palpable (Investigations) | 0 | 1 | 0
Thyroxine increased (Investigations) | 0 | 1 | 0
Tri-iodothyronine increased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Resting tremor (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract discomfort (Renal and urinary disorders) | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-06-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT02011945/SAP_000.pdf
  • Study Protocol (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT02011945/Prot_001.pdf